CLINICAL TRIAL: NCT03546023
Title: Assessment of Quality of Life in Patients With Chronic Cancer Pain Using Brief Pain Inventory. A Prospective Observational Study
Brief Title: Brief Pain Inventory to Assess Cancer Pain and Quality of Life
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Raghu Thota, Professor, Tata Memorial Hospital
Other Study IDs: 1921
Record Dates: First submitted 2018-03-26; First posted 2018-06-06 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Chronic Cancer Pain
Keywords: Chronic cancer pain; pain clinic; Brief Pain Inventory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient Interview — BPI scores will be asked by the Doctor or the Research Nurse

SUMMARY:
Cancer-related pain has a major adverse impact on functional status and quality of life. Recently, a Survey conducted in 2015 in 10 Asian countries showed that among cancer patients in Asian population, 86% of patients reported that their pain affected their activities of daily living, 87% their sleep, 92% their concentration and focus, and 67% excessive reliance on others. Only 34% reported a good quality of life. Effective pain management may help the patient to focus on the positive aspects of life, decreasing the focus on pain and also promote better adherence to reasonable treatment plans. Hence the emphasis is on improving the Quality of Life and not mere pain control.

DETAILED DESCRIPTION:
This is a Prospective Observational Study. All new patients in chronic pain OPD are been administered BPI questionnaire as a standard of practice in our institute, in the language best understood by them e.g. English, Hindi, Marathi, Bengali. The participants will be asked to complete it once during their first visit to the pain clinic, before the start of treatment or ongoing treatment for pain (Baseline) and then during subsequent visits (Follow up). Most chronic pain patients are advised to follow-up by one to two weeks. Patients who are willing to participate in the study will be included after obtaining an informed consent. Data will be collected from BPI, Chronic Pain Record form and EMR and will be analyzed. Demographic data, diagnosis, pain data sheet, drug treatment as well as other form of therapies will be recorded. There will be no direct communication with the patient and data of quality of life will be retrieved from pain clinic records.

The Brief Pain Inventory (BPI) long form and short form questionnaire is a validated multidimensional pain assessment tool developed by Cleeland and Ryan. It is one of the most commonly used measures for assessing both pain severity and interference with functions in adults with cancer, thereby satisfying two recommendations (assessment of pain to include both intensity and interference) set by the Initiative on Methods, Measurements, and Pain Assessment in Clinical Trials (IMMPACT) group. It is brief, self administered, easily understood and can be administered to large numbers of patients,.

It contains three questions regarding pain intensity and seven regarding pain interference that are rated on an ordinal numerical scale with anchors of 0 (no pain/interference) to 10 (maximum pain/interference). Pain intensity is measured according to the worst pain experienced in the last three days, average pain in the last three days, and current pain. Pain interference assesses how that pain has affected general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life. The sum of the scores of the pain intensity items represents the summed pain intensity score and the sum of the scores on the pain interference items represents the summed interference score. In addition, the patient enters his pain localization on a body drawing and can give details of his current medication.

ELIGIBILITY:
Inclusion Criteria:

* All patients registered in chronic pain OPD for 12 months from the date of approval of the study by IEC, at Tata Memorial Hospital.
* Age ≥ 18 years

Exclusion Criteria:

* Incomplete BPI forms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients attending the Pain Clinic over a period of 12 months aged 18 years and more.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Functional activity measurement using the Brief Pain Inventory (BPI) | followup visit (minimum 7 days)
  Any change in baseline score of functional activity from BPI during the followup visit.

CONTACTS AND LOCATIONS:
Overall Officials: Raghu Thota, MD, MNAMS, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No